CLINICAL TRIAL: NCT02189707
Title: Effects of 4-week Bifidobacterium-lactis HN019 Supplementation on Colonic Transit Time and Gastrointestinal Symptoms in Adults With Functional Constipation: A Double-blind, Randomized, Placebo-controlled Dose-ranging Trial
Brief Title: Effects of Probiotic Supplementation on Colonic Transit Time and Gastrointestinal Symptoms in Adults With Constipation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco Sweeteners Oy (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Bifido transit 3
Record Dates: First submitted 2014-07-04; First posted 2014-07-14 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Constipation; Gastrointestinal Disorder
Keywords: Gastrointestinal disorder; Constipation; Probiotics; Dietary supplement
MeSH Terms: conditions — Constipation; Gastrointestinal Diseases | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic Bifidobacterium 1x1010 cfu (Experimental): One capsule of study product, mixed with provided yogurt, will be consumed once a day.
  Interventions: Dietary Supplement: Probiotic Bifidobacterium 1x1010 cfu
- Probiotic Bifidobacterium 1x109 cfu (Experimental): One capsule of study product, mixed with provided yogurt, will be consumed once a day.
  Interventions: Dietary Supplement: Probiotic Bifidobacterium 1x109 cfu
- Placebo powder in capsules (Placebo Comparator): One capsule of study product, mixed with provided yogurt, will be consumed once a day.
  Interventions: Other: Placebo powder in capsules

INTERVENTIONS:
Dietary Supplement: Probiotic Bifidobacterium 1x1010 cfu — Participants who pass the initial screening will enter a 2-week placebo-only run-in period. Participants who successfully complete the run-in period will be randomized to daily supplementation with B. lactis HN019 (1 x 1010 cfu), B. lactis HN019 (1 x 109 cfu), or placebo for 4 weeks.
  Other Names: Probiotic powder (1 x1010 cfu B. lactis HN019) in capsules
  Arms: Probiotic Bifidobacterium 1x1010 cfu
Dietary Supplement: Probiotic Bifidobacterium 1x109 cfu — Participants who pass the initial screening will enter a 2-week placebo-only run-in period. Participants who successfully complete the run-in period will be randomized to daily supplementation with B. lactis HN019 (1 x 1010 cfu), B. lactis HN019 (1 x 109 cfu), or placebo for 4 weeks. One capsule of study product, mixed with provided yogurt, will be consumed once a day.
  Other Names: Probiotic powder (1 x 109 cfu B. lactis HN019) in capsules
  Arms: Probiotic Bifidobacterium 1x109 cfu
Other: Placebo powder in capsules — Participants will consume placebo capsules only during the 2-week run-in period. After randomization, participants will be administered their assigned study product and will continue on the product for 4 weeks.
  Arms: Placebo powder in capsules

SUMMARY:
To determine if Bifidobacterium lactis HN109 improves transit time and gastrointestinal symptoms in adults with constipation.

DETAILED DESCRIPTION:
Constipation is a commonly diagnosed gastrointestinal disorder with an estimated prevalence in the general population of 12-19%, which results in lower quality of life and significant healthcare costs to the individual. Almost 9 in 10 physician visits for constipation result in a laxative prescription. Additionally, consumers in the USA and in the United Kingdom spend almost 1 billion dollars annually for over-the-counter laxatives. Chronic constipation is diagnosed almost solely on patient symptoms, which generally includes unsatisfactory defecation due to infrequent stools, difficult stool passage, or both. The cause of chronic constipation is unknown and likely multifactorial with physiological changes, psychological factors, and lifestyle influences identified as possible culprits. Consequently, identification of effective constipation treatments remains a challenge.

The initial management of constipation symptoms is focused on evaluating lifestyle and diet variables as possible culprits. If lifestyle modifications are unsuccessful in alleviating constipation, various medications may be prescribed. In fact, about 50% of adults with constipation are not completely satisfied with available treatments. Consequently, there is a clear need for alternative constipation treatments that are safe, effective, and cost-effective.

Probiotics are live micro-organisms that result in a health benefit for the host when administered in adequate dosages. In recent years, probiotics have been commonly used to alleviate symptoms in a variety of gastrointestinal disorders. It is hypothesized that probiotics help to maintain gut lumen homeostasis by hindering growth of luminal pathogens and restoring the normal flora of the gut. As such, the use of probiotics for the relief of constipation symptoms is very promising. Numerous studies have been published addressing the utility of probiotics for gastrointestinal health including constipation. However, since probiotic efficacy is largely strain-specific, each specific strain must be individually tested in clinical trials.

Given the promising clinical results of probiotics on gastrointestinal health to date, the objective of this clinical trial is to evaluate the safety and effectiveness of 4-week Bifidobacterium lactis HN019 supplementation, in a dose-ranging fashion, on Colonic Transit Time (CTT) and gastrointestinal symptoms in adults with constipation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 70 years
* 2.Body mass index between 18.5 and 34.9 kg/m2
* 3. Meets the Rome III criteria for functional constipation as follows: (Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis):

  * Must meet 2 or more of the following criteria:

    * Straining during at least 25% of defecations
    * Lumpy or hard stools in at least 25% of defecations
    * Sensation of incomplete evacuation for at least 25% of defecations
    * Sensation of anorectal obstruction/blockage for at least 25% of defecations+ Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
    * Fewer than three defecations per week
  * Loose stools are rarely present without the use of laxatives
  * Insufficient criteria for irritable bowel syndrome

Exclusion Criteria:

* 1.Major gastrointestinal complication (e.g. Crohn's disease, ulcer)
* 2. Prior abdominal surgery that, in the opinion of the investigator, may present a risk for the participant or confound study results
* 3. Clinically significant underlying systemic illness that may preclude the participant's ability to complete the trial or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness)
* 4. Daily consumption of probiotics, prebiotics, fermented milk, and/or yogurt within 2 weeks of screening and throughout the trial other than the provided study products
* 5. Laxative use within 48 hours of screening (rescue medication allowed for intolerable symptoms during study)
* 6. Regular use of any drug or dietary supplement known to cause constipation (e.g. iron, opioids, sucralfate, misoprostol, 5-Hydroxytryptamine#-antagonists, antacids with magnesium, calcium or aluminum, antidiarrheal medication, anticholinergic agents, calcium supplements, calcium channel blockers, tricyclic antidepressants or nonsteroidal antiinflammatory drugs), within 1 month before screening.
* 7. Anticipated major dietary or exercise changes during the study
* 8. Systemic steroid use, within 1 month before screening.
* 9. Eating disorder
* 10. Contraindication to dairy products (e.g., intolerance to lactose or any substance in the study product)
* 11. History of alcohol, drug, or medication abuse
* 12. Pregnant or lactating female, or pregnancy planned during study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Colonic transit time | The primary outcome of Colonic Transit Time will be evaluated with abdominal x-rays on days 0 and 28

SECONDARY OUTCOMES:
Patient (syn. participant) assessment of constipation symptoms (PAC-SYM) | At days 0 and 28
Patient Assessment of Constipation Quality of Life (PAC-QoL) | At days 0 and 28
Bowel Function Index | At days 0 and 28
Adequate Relief of constipation (yes/no) | At days 0 and 28
Bowel movement frequency stools per week) | Participants will record the number of defecations per day in a daily diary during the 2-week run-in period and each day during the 4-week supplementation period
Stool consistency (Bristol Stool Scale) | Participants will record stool consistency during the 2-week run-in period and each day during the 4-week supplementation period.
Degree of Straining (1-5 scale) | Participants will record degree of straining during the 2-week run-in period and each day during the 4-week supplementation period.
Participant assessment of bowel emptying (yes/no) | Participants will record sensation of complete bowel emptying during the 2-week run-in period and each day during the 4-week supplementation period.
Abdominal discomfort/bloating (1-5 scale) | Participants will record severity of abdominal discomfort and bloating during the 2-week run-in period and each day during the 4-week supplementation period.
Overall product satisfaction (1-5 scale) | At the end of the supplementation period (D28)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Latreille-Barbier, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- EUROFINS OPTIMED Clinical Research, Gières, France